CLINICAL TRIAL: NCT05008146
Title: Imaging Corticotrophin-releasing Factor (CRF) X Nociceptive Opioid Peptide (NOP) Interactions in Cocaine Use Disorders (Aim 1)
Brief Title: Imaging CRF X NOP Interactions in CUD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rajesh Narendran (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Rajesh Narendran, Professor of Radiology and Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20060171 (Aim 1); R01DA026472 (NIH); STUDY19110156 (Other: University of Pittsburgh)
Record Dates: First submitted 2021-08-11; First posted 2021-08-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine use disorder; [C-11]NOP-1A PET; Nociceptive opioid peptide receptors
MeSH Terms: interventions — BaseLine dental cement; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Cocaine Use disorder and Healthy control groups will receive same interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET (Experimental): [C-11]NOP-1A
  Interventions: Radiation: Baseline [C-11]NOP-1A PET Scan; Drug: Hydrocortisone; Radiation: Post-hydrocortisone [C-11]NOP-1A PET Scan

INTERVENTIONS:
Radiation: Baseline [C-11]NOP-1A PET Scan — Radiotracer
Drug: Hydrocortisone — Intravenous, 1mg/Kg
Radiation: Post-hydrocortisone [C-11]NOP-1A PET Scan — Radiotracer

SUMMARY:
This study uses [11C]NOP-1A positron emission tomography (PET) and a hydrocortisone challenge to image the interaction between nociceptive opioid peptide (NOP) receptors and cortisol/corticotrophin releasing factor (CRF) in subjects with cocaine use disorders (CUD) and matched healthy controls (HC). It will also examine whether alterations in CRF x NOP interactions predict relapse in subjects with CUD.

DETAILED DESCRIPTION:
Cocaine use disorder (CUD) is a chronic disorder associated with numerous relapses and periods of abstinence.

Studies in CUD suggest that ~ 60 to 75% of abstinent addicts relapse over twelve months Documenting specific neurochemical abnormalities that lead to relapse in individuals with CUD has the potential to accelerate the development of medications to prevent relapse. Basic investigations postulate an imbalance between brain stress and anti-stress/resilience systems as the underlying mechanism that drives negative reinforcement, craving, and relapse in addiction. Nociceptin (N/OFQ), which binds to the nociceptive opioid peptide receptors (NOP) is a critical component of the brain's anti-stress system. N/OFQ counteracts the functional effects of the primary stress-promoting neuropeptide corticotrophin releasing factor (CRF) in the brain to exert its anti-stress effects. Studies have also shown that acute increases in CRF and stress are countered by increased NOP receptor expression (~ 10% ) in brain regions that regulate stress such as bed nucleus of the stria terminalis. PET studies with the NOP radiotracer [11C]NOP-1A show increased binding to NOP in CUD compared to HC. PET studies also show NOP receptors to upregulate (~ 15%) in response to an acute intravenous hydrocortisone challenge (1 mg/Kg). NOP upregulation may represent an adaptive mechanism in the brain to counteract stress-induced increases in cortisol and CRF. Here, we postulate a failure in this adaptive mechanism as a reason that leads to relapse in CUD. CUD subjects and HC will be studied with [11C]NOP-1A before and after an intravenous hydrocortisone challenge (aim 1). Hydrocortisone is used as a challenge because it increases cortisol and CRF in brain regions that regulate stress. We hypothesize that hydrocortisone-induced increases in [11C]NOP-1A binding (DELTA VT) will be smaller in CUD relative to HC, and this will be associated with less time to relapse in a 12-week follow up.

ELIGIBILITY:
Cocaine use disorders (CUD)

1. Males or females between 18 and 55 years old
2. Fulfil DSM-5 criteria for cocaine use disorder
3. No other current DSM-5 psychiatric or addictive disorders (such as major depressive disorder, bipolar disorders, psychotic disorders, etc.,)
4. No current abuse (six months) of opiates, sedative-hypnotics, amphetamines, MDMA, etc., as well as moderate to severe alcohol or cannabis use (twice a week). Nicotine use will be quantified and controlled between groups using the Fagerstrom Test for Nicotine Dependence (Heatherton et al., 1991);
5. Not currently on prescription medical or psychotropic medications
6. No current or past severe medical, endocrine or neurological illnesses including glaucoma, seizure disorders, hypertension, hypercholesterolemia as assessed by a complete medical history and physical
7. Not currently pregnant or breastfeeding
8. No history of significant radioactivity exposure in past year from another research study or occupation that exceeds RDRC guidelines
9. No metallic objects in the body that are contraindicated for MRI

Healthy Controls (HC)

1. Males or females between 18 and 55 years old
2. No present or past DSM-5 disorders (other than nicotine dependence)
3. Criteria 5 to 9 as listed previously.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
DELTA VT | Baseline, and 3 hours post-hydrocortisone
  VT is the volumes of distribution expressed relative to total plasma ligand concentration; Delta VT is the change in VT from baseline to 3-hours post-hydrocortisone.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Narendran, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No